CLINICAL TRIAL: NCT02446158
Title: A Randomized Trial of Daily Chlorhexidine Care at the Exit Site in Peritoneal Dialysis Patients for Bacterial Decolonization and Prevention of Infection
Brief Title: Daily Chlorhexidine Care at the Exit Site in Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EDAHP99020
Record Dates: First submitted 2015-05-10; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Peritoneal Dialysis Catheter Exit Site Infection
MeSH Terms: interventions — chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorhexidine gluconate (Experimental): PD (peritoneal dialysis) paitents with daily chlorhexidine exit site care
  Interventions: Drug: Chlorhexidine gluconate
- Control group (No Intervention): PD (peritoneal dialysis) patients with usual (Normal saline) exit site care

INTERVENTIONS:
Drug: Chlorhexidine gluconate — The intervention group received daily cleaning of the exit site and application of 4% chlorhexidine (Antigerm Solution, Shining BioMedical Com. Ltd) with a swab. The chlorhexidine was rinsed off after 3 min of air drying and then gauze was applied.
  Other Names: Chlorhexidine
  Arms: Chlorhexidine gluconate

SUMMARY:
Chlorhexidine is used in central line dressing changes and is effective in reducing line infections. It is unclear if daily chlorhexidine care at the exit site in peritoneal dialysis (PD) patients can reduce the risk of Staphylococcus aureus (SA) colonization or exit site infection.

DETAILED DESCRIPTION:
There is no consensus on what regimen is optimal for topical care of the peritoneal dialysis (PD) catheter exit site. Several methods including soap and water, povidone-iodine, hydrogen peroxide, chlorhexidine, and topical antimicrobial agents such as gentamicin or mupirocin cream have been described for care of the exit site. However, many of these studies were small or short-term and lacked longitudinal evaluation of bacterial decolonization efficacy. Staphylococcus aureus (SA) is one of most common causes of peritonitis and exit-site infection and is associated with a high PD catheter removal rate. Carriers of SA had a higher rate of exit-site infection than non-carriers. In previous studies, staphylococcal carriage prophylaxis using either mupirocin or gentimicin ointment in the nares or exit site significantly reduced the rate of exit-site infection due to SA. However, emerging antibiotic resistance is a concern. In addition, MRSA infection in PD patients is more severe than other pathogens; therefore, choosing a good antiseptic for SA and/or MRSA decolonization is important.

In recent years, the use of chlorhexidine in bathing or central line dressing changes was implemented to prevent bacterial colonization and multidrug resistant bacterial infections and was also used in hemodialysis patients. Data regarding chlorhexidine used in the catheter care of PD patients are limited and it is unclear if the use of chlorhexidine for exit site care contributes to long-term bacterial decolonization and acts as a prophylaxis for exit site infections.

ELIGIBILITY:
Inclusion Criteria:

* patients > 20 years old who received PD for more than 3 months

Exclusion Criteria:

* a history of psychological illness or condition that interferes with caring of a wound
* recent (within 1 month) exit-site infection, peritonitis, or tunnel infection
* recent treatment with an antibiotic administered by any route in the last month
* or known hypersensitivity to or intolerance of chlorhexidine or mupirocin

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
exit site bacterial colonization status | 1 year
  We performed swab cultures at the exit site and nasal site every month during follow-up at the hospital and analyzed the bacterial colonization status at 6 and 12 months as the primary outcome.

SECONDARY OUTCOMES:
The exit-site infection rate | 1 year
  An exit-site infection was defined by the presence of purulent drainage, with or without erythema of the skin at the catheter-epidermal interface.

REFERENCES:
- [Derived] Wang HH, Hung SY, Chang MY, Lee YC, Lin HF, Lin TM, Yang SP, Lin HH, Yang SC, Wang JL. Bacterial colonization patterns in daily chlorhexidine care at the exit site in peritoneal dialysis patients-A prospective, randomized controlled trial. PLoS One. 2017 Oct 5;12(10):e0184859. doi: 10.1371/journal.pone.0184859. eCollection 2017. PMID 28981543